CLINICAL TRIAL: NCT06317441
Title: The Safety And Efficacy Of A Probiotic Intervention On Lactulose Hydrogen Breath Test-Positive Patients And Related Gastrointestinal Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nimble Science Ltd. (Industry)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIMCSF137
Record Dates: First submitted 2024-02-27; First posted 2024-03-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Small Intestinal Bacterial Overgrowth; SIBO
Keywords: Functional abdominal bloating and distension; Functional Diarrhea; Irritable Bowel Syndrome with Diarrhea; Irritable Bowel Syndrome; Abdominal Bloating; IBS; IBS-D; FABD; Functional Gastrointestinal Disorders; FGID
MeSH Terms: conditions — Dilatation, Pathologic; Irritable Bowel Syndrome; Gastrointestinal Diseases | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Probiotic (High dose) (Experimental): A high dosage probiotic per capsule
  Interventions: Dietary Supplement: Probiotic
- Probiotic (Low dose) (Experimental): A low dosage probiotic per capsule
  Interventions: Dietary Supplement: Probiotic
- Control group (Placebo) (No Intervention): No probiotic dosage

INTERVENTIONS:
Dietary Supplement: Probiotic — The intervention consists of a probiotic either with a low or high dosage
  Arms: Probiotic (High dose); Probiotic (Low dose)

SUMMARY:
The goal of this study is to test the effect of a probiotic formulation on gastrointestinal symptoms, gut and small intestine microbiota in participants suffering from small intestinal bacterial overgrowth (SIBO). Two doses of probiotic will be evaluated against placebo.

DETAILED DESCRIPTION:
The goal of this double-blinded, randomized, placebo-controlled clinical study is to evaluate whether two different doses of a probiotic formulation may have effect on gastrointestinal symptoms, as well as gut and small intestine microbiota, in participats suffering from SIBO. The two probiotic doses will be compared to a placebo.

The main research questions to be answered by this study are related to:

* Probiotic effect on bloating and abdominal distension.
* Probiotic effect on other gastrointestinal symptoms.
* Probiotic effect on incidence of SIBO.
* Probiotic effect on small intestine and gut microbiota.

The study will include a 2 month intervention with the investigational products and assessments will be conducted at baseline, mid-intervention, end-of-intervention, and follow-up period, with the exception of SIBO diagnosis, which will be conducted at baseline and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years old at the inclusion of the study, both female and male subjects.
2. Signed Informed Consent; willing and able to comply with study procedures.
3. Willing to maintain their diet and physical activity levels during the study.
4. Able to swallow a size-00 capsule (23mm length and 9mm width).
5. Participants with at least one of the following Rome IV diagnoses: FABD, functional diarrhea, IBS-M, or IBS-D.
6. Baseline weekly average of worst daily (in past 24 hours) abdominal bloating/distension score of >= 3.0 on a 0-to-10-point scale.
7. Participants with abnormal LHBT following the North American Consensus recommendations (A rise in hydrogen of ≥20 ppm by 90 min).

Exclusion Criteria:

1. History of less than three (3) bowel movements per week.
2. With the diagnosis of IBS-C.
3. Prior gastrointestinal disease, surgery, or abdominal or pelvic radiation treatment which, in the Investigator's opinion, would lead to intestinal structuring or obstruction with a risk of capsule non-excretion, including, e.g., achalasia, eosinophilic esophagitis, any IBD, or previous esophageal, gastric, small intestinal, or colonic surgery. Appendectomy or cholecystectomy more than 3 months before the screening visit is acceptable.
4. Persons with central venous catheters.
5. History of known structural gastrointestinal abnormalities such as structures or fistulas leading to mechanical obstruction.
6. Known history abdominal radiation treatment.
7. Use of any medications in the week prior to the screening study visit, unless part of regular treatment, that could substantially alter gastrointestinal motor function (e.g., opioids, anticholinergics, or GLP-1 analogues); laxative use is allowed if used less than 3 times a week and it is willing to keep unchanged in the week prior to the SIMBA capsule ingestions. Proton pump inhibitors (PPIs) are allowed provided a wash-out period of 48 hours is respected before swallowing the SIMBA capsules and PPI treatment is resumed only 4 hours thereafter.

   o Prokinetic use. Potential participants who are not using prokinetics to treat SIBO may be eligible after a 2-week washout period, and willing to not use prokinetics for the study duration.
8. Unable to stop using laxatives or prokinetic medications for 4 days before the study procedure (BT). Laxatives can be resumed after the test is conducted.
9. Organic motility disorder, including gastroparesis, intestinal pseudo-obstruction, systemic sclerosis, Ogilvie's syndrome.
10. Celiac disease (treated or untreated).
11. Any significant heart, liver, lung, kidney, blood, endocrine or nervous system disease, which in the opinion of the investigator, would adversely affect study safety or outcome.
12. Cancer diagnosis or treatment within the past year (non-melanoma skin cancers are acceptable).
13. Gastrointestinal inflammatory diseases, including ulcerative colitis, Crohn's disease, microscopic colitis.
14. Participants with IBS presenting with alarm symptoms such as: rectal bleeding, unexplained weight loss, iron deficiency anemia, and nocturnal symptoms,
15. Participants over the age of 50 or older who have not had:

    * a colon cancer screening by either a negative FIT or FOBT test within the last 2 years; OR
    * a colonoscopy in the prior 10 years which was negative for colorectal cancer
16. Epilepsy diagnosis.
17. History or diagnosis of immunological diseases, infectious diseases or immune-compromised conditions, which in the opinion of the investigator, would adversely affect study safety or outcome. Such as, but not limited to, hepatitis, tuberculosis, HIV positive, Parkinson's, multiple sclerosis, AIDS, lymphoma, and long-term corticosteroid treatment.
18. History of oropharyngeal dysphagia, or other swallowing disorder with a risk of capsule aspiration.
19. Antibiotic use (except for topical use) ≤ 12 weeks prior to screening. Potential participants may be eligible once a 12-week washout is completed.
20. Regular use of probiotics, prebiotics or synbiotics (including food and drinks containing added probiotics and/or probiotic yogurts with live, active cultures) within 1 month prior to screening. Potential participants may be eligible once a 1-month washout is completed.
21. Any prior Fecal Microbiota Transplantation.
22. Pregnant or breastfeeding.
23. Planning to become pregnant.
24. Alcohol or drug abuse.
25. Allergy to the components present in the probiotic and placebo capsules.
26. Are non-English speaking.
27. Are scheduled for an MRI at any time during the study. Potential participants may be eligible to participate once their MRI procedure is completed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in bloating/distension severity | From baseline to end of intervention (week 8).
  The primary outcome will assess the changes in weekly median severity of bloating/distension, defined as pressure, fullness or sensation of increased girth with a daily assessment with an ordinal scale between probiotic groups and placebo.

SECONDARY OUTCOMES:
Median bloating-free days | Each intervention week and follow up (week 12) compared to baseline.
  Median bloating-free days per week at each intervention week and follow up
Change in median bloating/distension severity | At all intervention weeks (with the exception of end-of-intervention, as described in the primary outcome) and follow-up (week 12) compared to baseline.
  Change in median bloating/distension severity assessed by an ordinal scale (0 no severity- 10 extreme severity) at all intervention weeks (with the exception of end-of-intervention, as described in the primary outcome)
Change in abdominal discomfort/pain | At mid-intervention (week 4), end of intervention (week 8), and follow-up (week 12) compared to baseline
  Change in abdominal discomfort/pain assessed by an ordinal scale (0 no pain - 10 extreme pain)
Changes in gastrointestinal symptoms | At mid-intervention (week 4), end of intervention (week 8), and follow-up (week 12) compared to baseline.
  Changes in gastrointestinal symptoms assessed with GSRS
Changes in stool frequency and consistency | At mid-intervention (week 4), end of intervention (week 8), and follow-up (week 12) compared to baseline.
  Changes in stool frequency and consistency assessed with the Bristol Stool Scale (scoring 1 watery - 7 hard)
Changes in the quality of life | At mid-intervention (week 4), end of intervention (week 8), and follow-up (week 12) compared to baseline.
  Changes in the quality of life assessed with the Short Form (SF)-36 questionnaire
Changes in reflux incidence and severity | At mid-intervention (week 4), end of intervention (week 8), and follow-up (week 12) compared to baseline.
  Changes in reflux incidence and severity assessed with the modified reflux symptoms (mRESQ)
Changes in the severity of IBS symptoms | At mid-intervention (week 4), end of intervention (week 8), and follow-up (week 12) compared to baseline.
  Changes in the severity of IBS symptoms assessed with IBS Severity Scoring System (IBS-SSS) questionnaire
Recovery rate of the probiotic strain | At mid-intervention (week 4) end of intervention (week 8), and follow-up (week 12) compared to baseline.
  Recovery rate of the probiotic strain in small intestine and stool specimens
Microbiome changes within small intestine, fecal and saliva samples | At mid-intervention (week 4), end of intervention (week 8), and follow-up (week 12) compared to baseline.
  Changes in the the bacterial populations with the small intestine, fecal and saliva microbiomes represented as a diversity ratio
Investigation how the microbiome and SIBO associate with each other though bacterial population analyses. | Through study completion, an average of 1 year
  Exploring the correlation of select bacterial populations with SIBO through analysis of the small intestine and fecal microbiomes using metagenomics methodologies.
Change in SIBO positivity rate | Through study completion, an average of 1 year
  Change in SIBO positivity rate assessed by glucose breath test

OTHER OUTCOMES:
Exploratory metabolomic analysis | Through study completion, an average of 1 year
  To investigate whether certain metabolites present in the small intestine, fecal, saliva samples may be associated with the presence/absence of SIBO. Using untargeted metabolomic methodologies.
Exploratory: Quantifying the probiotic cell proportions | Through study completion, an average of 1 year
  Determine the proportion of probiotic cells in spore versus germinated form using qPCR methodologies
Safety outcomes | Through study completion, an average of 1 year
  To collect safety data on the probiotic formulation and the SIMBA capsule by monitoring adverse events throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Nimble Science, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Select data with be shared with the participants